CLINICAL TRIAL: NCT00710580
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Comparing the Efficacy and Safety of ABT-874 to Etanercept and Placebo in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Study Comparing the Efficacy and Safety of ABT-874 to Etanercept and Placebo in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Paragon Biomedical (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M10-315
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Moderate to Severe Plaque Psoriasis
MeSH Terms: interventions — briakinumab; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Biological: ABT-874
- B (Active Comparator)
  Interventions: Biological: etanercept
- C (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: ABT-874 — SQ injection 200 mg Weeks 0 and 4; 100 mg Week 8
  Arms: A
Biological: etanercept — SQ injection 50 mg BIW
  Arms: B
Drug: placebo — SQ placebo injections for ABT-874 and etanercept
  Arms: C

SUMMARY:
Compare the efficacy of ABT-874 versus etanercept in subjects with moderate to severe plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Psoriasis for 6 MO
* BSA 10%
* PASI 12 or above
* PGA 3 or above

Exclusion Criteria:

* Previous exposure to either etanercept or ABT-874

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a PGA of 0 or 1 response relative to baseline at Week 12 | 12 Weeks
Proportion of subjects who achieve a PASI 75 response relative to baseline at Week 12 | 12 Weeks

SECONDARY OUTCOMES:
Proportion of subjects who achieve a PASI 100 response relative to baseline at Week 12 | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaul, MD, Study Director — AbbVie
Locations (42):
- United States (42):
  - Site Reference ID/Investigator# 9984, Birmingham, Alabama
  - Site Reference ID/Investigator# 10605, Birmingham, Alabama
  - Site Reference ID/Investigator# 10001, Scottsdale, Arizona
  - Site Reference ID/Investigator# 10502, Little Rock, Arkansas
  - Site Reference ID/Investigator# 9985, Bakersfield, California
  - Site Reference ID/Investigator# 10661, Irvine, California
  - Site Reference ID/Investigator# 14701, Los Angeles, California
  - Site Reference ID/Investigator# 9785, San Diego, California
  - Site Reference ID/Investigator# 10662, Santa Monica, California
  - Site Reference ID/Investigator# 10642, Vallejo, California
  - Site Reference ID/Investigator# 10263, New Haven, Connecticut
  - Site Reference ID/Investigator# 10503, Jacksonville, Florida
  - Site Reference ID/Investigator# 10266, Miami, Florida
  - Site Reference ID/Investigator# 9901, Miami, Florida
  - Site Reference ID/Investigator# 10501, West Palm Beach, Florida
  - Site Reference ID/Investigator# 15201, Alpharetta, Georgia
  - Site Reference ID/Investigator# 10762, Atlanta, Georgia
  - Site Reference ID/Investigator# 10262, Newnan, Georgia
  - Site Reference ID/Investigator# 9789, Snellville, Georgia
  - Site Reference ID/Investigator# 10666, Maywood, Illinois
  - Site Reference ID/Investigator# 15142, Plainfield, Indiana
  - Site Reference ID/Investigator# 10265, Louisville, Kentucky
  - Site Reference ID/Investigator# 15750, Owensboro, Kentucky
  - Site Reference ID/Investigator# 9790, Owensboro, Kentucky
  - Site Reference ID/Investigator# 9788, Fort Gratiot, Michigan
  - Site Reference ID/Investigator# 10604, Grand Blanc, Michigan
  - Site Reference ID/Investigator# 10541, Fridley, Minnesota
  - Site Reference ID/Investigator# 10641, St Louis, Missouri
  - Site Reference ID/Investigator# 10606, Omaha, Nebraska
  - Site Reference ID/Investigator# 10644, Omaha, Nebraska
  - Site Reference ID/Investigator# 9786, Berlin, New Jersey
  - Site Reference ID/Investigator# 10241, New York, New York
  - Site Reference ID/Investigator# 9787, Rochester, New York
  - Site Reference ID/Investigator# 9902, Hickory, North Carolina
  - Site Reference ID/Investigator# 10581, Wilmington, North Carolina
  - Site Reference ID/Investigator# 10504, Dayton, Ohio
  - Site Reference ID/Investigator# 10643, Knoxville, Tennessee
  - Site Reference ID/Investigator# 9981, Dallas, Texas
  - Site Reference ID/Investigator# 10264, San Antonio, Texas
  - Site Reference ID/Investigator# 9982, Webster, Texas
  - Site Reference ID/Investigator# 10182, Seattle, Washington
  - Site Reference ID/Investigator# 10321, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Strober BE, Crowley JJ, Yamauchi PS, Olds M, Williams DA. Efficacy and safety results from a phase III, randomized controlled trial comparing the safety and efficacy of briakinumab with etanercept and placebo in patients with moderate to severe chronic plaque psoriasis. Br J Dermatol. 2011 Sep;165(3):661-8. doi: 10.1111/j.1365-2133.2011.10419.x. Epub 2011 Jul 28. PMID 21574984